CLINICAL TRIAL: NCT06666517
Title: The Relationship Between the Density of Cancer-Associated Fibroblasts in the Peritumoral Stroma and Clinicopathological Data in Breast Cancer Patients
Acronym: PERICAFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Dogukan Akkus, Principal Investigator, Haydarpasa Numune Training and Research Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: HNEAH-GAEK 2024/149; Unit of Scientific Research (Other: University of Health Sciences)
Record Dates: First submitted 2024-10-08; First posted 2024-10-30 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Breast Carcinoma
Keywords: cancer associated fibroblast; breast cancer; tumor microenvironment
MeSH Terms: conditions — Breast Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- 1- Subtyping of Breast Cancer Patients. (Sham Comparator): Biopsy collection from patients who were diagnosed with breast cancer, subtyping of biopsy materials, and identification of patients with Luminal A, Luminal B, HER2 positive group, and triple-negative types.
  Interventions: Other: Immunohistochemistry Analysis
- 5- Surgery Phase (Sham Comparator): Surgery after neoadjuvant chemotherapy
  Interventions: Procedure: surgery (any volume) and / or pharmaceuticals treatment initiated or planned or only dynamic observation, in accordance with current clinical guidelines
- 2- Identification of patients to be included in the study. (No Intervention): Identification of patients diagnosed with breast cancer who meet the study's eligibility criteria.
- 3- Second Biopsy (Experimental): Taking biopsies from the center of the tumor and the peritumoral stroma of the same mass during marking of the mass before neoadjuvant chemotherapy
  Interventions: Procedure: Second Biopsy
- 4- Detection of cancer-associated fibroblasts (No Intervention): Analysis of cancer-associated fibroblasts using immunohistochemical methods on materials taken from the periphery and center of patients' tumors during the second biopsy.
- 6- Statistically Analyze (No Intervention): The investigators compare cancer-associated fibroblast densities by analyzing monitored patients' clinical and pathological data and statistically analyze and interpret the results.

INTERVENTIONS:
Procedure: surgery (any volume) and / or pharmaceuticals treatment initiated or planned or only dynamic observation, in accordance with current clinical guidelines — Routine surgery after neoadjuvant chemotherapy for breast cancer according to current guidelines.
  Arms: 5- Surgery Phase
Other: Immunohistochemistry Analysis — Determination of breast cancer subtypes through immunohistochemical analysis, and selection of Luminal B, HER2-positive, and triple-negative groups.
  Arms: 1- Subtyping of Breast Cancer Patients.
Procedure: Second Biopsy — Taking biopsies from the center of the tumor and the peritumoral stroma of the same mass during marking of the mass before neoadjuvant chemotherapy
  Arms: 3- Second Biopsy

SUMMARY:
Research Question:

Is there a relationship between the clinical prognosis and pathological data of breast cancer patients and the density of cancer-associated fibroblasts in the peritumoral stroma?

Objectives of the Study:

1. Detection of cancer-associated fibroblasts in the tumor microenvironment across different breast cancer subtypes.
2. Examination of the correlation between the clinical prognosis and pathological data of patients with different breast cancer subtypes and cancer-associated fibroblast subtypes.

The goal of this study based on the correlation obtained, the aim is to propose cancer-associated fibroblasts as a more effective marker for breast cancer classification and prognosis.

DETAILED DESCRIPTION:
During the routine marking before neoadjuvant chemotherapy of breast cancer patients with triple-negative, HER2-positive, or Luminal B molecular subtypes, the correlation between the density of cancer-associated fibroblasts in the samples taken from the center of the tumor and the peritumoral stroma of the same mass with the patient's clinical prognosis and pathological data will be examined.

Approach and Methods:

Collection of Tissue Samples via Core Needle Biopsy from Breast Cancer Patients (Luminal B, HER2 Group, and Triple-Negative Group):

Breast masses will be examined supine using an ultrasound machine with a 14 MHz linear transducer. The tumor and peritumoral parenchyma will be evaluated using a 1.5 T MRI machine with a 16-channel breast coil, in the prone position, under dynamic contrast-enhanced and diffusion-weighted imaging guidance. Under sonographic guidance and local anesthesia, one tissue sample will be taken from the center of the mass using a 14G/10 cm core needle immediately before marking for neoadjuvant chemotherapy. One tissue sample will be taken from the peritumoral stroma where diffusion restriction is shown in diffusion-weighted MRI from patients diagnosed with Luminal B, HER2, or triple-negative malignancy.

Identification of Cancer-Associated Fibroblasts via Immunohistochemical Analysis:

For immunohistochemical analysis, 3 µm thick sections will be taken from paraffin blocks prepared from the core needle biopsy tissues from the periphery of the tumor, and the blocks will be deparaffinized in an incubator at 60 °C. The prepared slides will be stained using the LEICA Bond III fully automated IHC system, with the FAPα antibody, SMA antibody, and PDGFR-β antibody. Diaminobenzidine (DAB) will be used as the chromogen. Positive control tissues will include Fibroblast Activation Protein, alpha [SP325] Conc. 0.1mL (1:100) colon adenocarcinoma, Actin Smooth Muscle [1A4] Conc. 0.1mL (1:100-500) appendix, and PDGFR-B [D-6] C.Liq.1ml (1:50-500) kidney.

The immunohistochemical analysis of the patient under clinical follow-up will be compared with the type of surgery performed, the pathological data, and the clinical prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with histopathologically confirmed Luminal B, HER2-positive, or triple-negative breast cancer subtypes.
* Patients who have not previously received any neoadjuvant chemoradiotherapy.
* Patients over 18 years of age.
* Adequate cellularity in biopsies obtained via core needle biopsy.

Exclusion Criteria:

* Patients diagnosed with histopathologically confirmed Luminal A breast cancer subtype.
* Patients who have previously received any neoadjuvant chemoradiotherapy.
* Patients under 18 years of age.
* Inadequate cellularity in biopsies obtained via core needle biopsy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study aims to detect cancer-associated fibroblasts in female breast cancer. Male breast cancer has a different mechanism from female breast cancer.
Enrollment: 69 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Detection of Cancer-Associated Fibroblasts via Immunohistochemical Analysis | Within 4 weeks after immunohistochemical staining.
  The detection of cancer-associated fibroblasts will be conducted separately using each immunohistochemical stain, and after the density(percentage) and intensity(will be scored 1 to 4) are assessed, the H-score(percentage X intensity score) will be determined by an expert pathologist, followed by grouping.

SECONDARY OUTCOMES:
Collecting Patient Information From The Hospital System | Within 1 year after surgery
  Patients who underwent surgery after neoadjuvant chemotherapy will be monitored based on the following parameters in the pathology specimen: estrogen receptor(positive or negative), progesterone receptor(positive or negative), HER2 receptor(positive or negative), percentage of Ki67, nuclear grade(1,2 or 3), tumor diameter in centimeters, percentage of tumor-infiltrating lymphocytes, presence of in situ carcinoma, presence of multifocality, presence of lymphovascular invasion, residual cancer burden score(MD Anderson RCB Score) and clinically performed axillary and breast surgeries(breast sparing mastectomy, skin sparing mastectomy, nipple sparing mastectomy, modified radical mastectomy, axillary dissection or sentinel lymph node dissection), presence of recurrence and metastasis, whether they underwent reoperation, overall and disease-free survival in days and presence of mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Meryem Gunay Gurleyik, Medical Doctor, Study Director — Haydarpasa Numune Training and Research Hsopital
Locations (1):
- Haydarpasa Numune Training and Research Hospital, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Everything can be accessible.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After August 2025 the investigators will share the information and there will be no end date.
Access Criteria: Everyone affiliated academically can access it.

REFERENCES:
- [Background] Giorello MB, Borzone FR, Labovsky V, Piccioni FV, Chasseing NA. Cancer-Associated Fibroblasts in the Breast Tumor Microenvironment. J Mammary Gland Biol Neoplasia. 2021 Jun;26(2):135-155. doi: 10.1007/s10911-020-09475-y. Epub 2021 Jan 4. PMID 33398516
- [Background] Barriga V, Kuol N, Nurgali K, Apostolopoulos V. The Complex Interaction between the Tumor Micro-Environment and Immune Checkpoints in Breast Cancer. Cancers (Basel). 2019 Aug 19;11(8):1205. doi: 10.3390/cancers11081205. PMID 31430935
- [Background] Wall SW, Echeverria GV. Avoiding Extinction: Cancer-Associated Fibroblasts Help Triple-Negative Breast Cancer Outrun Chemotherapy. Cancer Res. 2023 Nov 15;83(22):3667-3669. doi: 10.1158/0008-5472.CAN-23-2770. PMID 37964615
- [Background] Benyahia Z, Dussault N, Cayol M, Sigaud R, Berenguer-Daize C, Delfino C, Tounsi A, Garcia S, Martin PM, Mabrouk K, Ouafik L. Stromal fibroblasts present in breast carcinomas promote tumor growth and angiogenesis through adrenomedullin secretion. Oncotarget. 2017 Feb 28;8(9):15744-15762. doi: 10.18632/oncotarget.14999. PMID 28178651
- [Background] Eiro N, Gonzalez LO, Fraile M, Cid S, Schneider J, Vizoso FJ. Breast Cancer Tumor Stroma: Cellular Components, Phenotypic Heterogeneity, Intercellular Communication, Prognostic Implications and Therapeutic Opportunities. Cancers (Basel). 2019 May 13;11(5):664. doi: 10.3390/cancers11050664. PMID 31086100
- [Background] Salimifard S, Masjedi A, Hojjat-Farsangi M, Ghalamfarsa G, Irandoust M, Azizi G, Mohammadi H, Keramati MR, Jadidi-Niaragh F. Cancer associated fibroblasts as novel promising therapeutic targets in breast cancer. Pathol Res Pract. 2020 May;216(5):152915. doi: 10.1016/j.prp.2020.152915. Epub 2020 Mar 2. PMID 32146002
- [Background] Pelon F, Bourachot B, Kieffer Y, Magagna I, Mermet-Meillon F, Bonnet I, Costa A, Givel AM, Attieh Y, Barbazan J, Bonneau C, Fuhrmann L, Descroix S, Vignjevic D, Silberzan P, Parrini MC, Vincent-Salomon A, Mechta-Grigoriou F. Cancer-associated fibroblast heterogeneity in axillary lymph nodes drives metastases in breast cancer through complementary mechanisms. Nat Commun. 2020 Jan 21;11(1):404. doi: 10.1038/s41467-019-14134-w. PMID 31964880